CLINICAL TRIAL: NCT02009800
Title: ICI-VPH: Impact Des Calendriers d'Immunisation Contre Les HPV
Brief Title: ICI-VPH: Impact of HPV Immunisation Schedules Against HPV
Acronym: ICI-VPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other); Ministere de la Sante et des Services Sociaux (Other); Institut National en Santé Publique du Québec (Other)
Responsible Party: Principal Investigator, Chantal Sauvageau, Co-principal investigator, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ICI-VPH-1
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Human Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 dose of quadrivalent HPV vaccine (No Intervention): The participants who have already received 2 doses of the quadrivalent HPV vaccine (0, 6 months schedule) 5 years before recruitment will not receive an additional dose.
- 3 doses of quadrivalent HPV vaccine (Experimental): The participants will receive a 3rd dose of quadrivalent HPV vaccine at recruitment visit, which is 5 years after having received two doses of vaccine given 6 months apart in grade 4 (0, 6, 60 months Schedule)
  Interventions: Biological: Quadrivalent HPV vaccine

INTERVENTIONS:
Biological: Quadrivalent HPV vaccine — One dose of Gardasil administered in the intervention group
  Other Names: Gardasil
  Arms: 3 doses of quadrivalent HPV vaccine

SUMMARY:
This randomised clinical trial aims to determine whether an immunization schedule comprising two doses of Gardasil administered six months apart is non-inferior to a schedule comprising three doses administered at 0, 6 and 60 months for the prevention of HPV-16 and HPV-18 infections that persist for at least six months, up to ten years after the initial vaccination.

The study hypothesis is that the two-dose schedule would offer similar protection as that of a three-dose schedule against persistent HPV-16/18 infections.

ELIGIBILITY:
Inclusion Criteria:

* Having received two doses of Gardasil in 2008-2009, 2009-2010,2010-2011 or 2011-2012 according to 0, 6 months Schedule (between 4 and 12 months)
* Resident of the regions chosen for the study

Exclusion Criteria:

* Being considered immunosuppressed at time of vaccination (9-10 years-old) or at recruitment visit
* Being pregnant at recruitment visit

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3364 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Incidence of persistent HPV-16/18 infections | 5 years after recruitment visite

SECONDARY OUTCOMES:
Geometric mean titres of antibodies and seropositivity for HPV types 6, 11, 16 and 18 | 5 years after recruitment visit

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre Hospitalier Uiversitaire de Montréal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec, CHU de Québec, Québec

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Sauvageau C, Mayrand MH, Ouakki M, Ionescu IG, Coutlee F, Lacaille J, Benoit M, Gilca V. Protection Against Persistent HPV-16/18 Infection After Different Number of Doses of Quadrivalent Vaccine in Girls and Young Women: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2519095. doi: 10.1001/jamanetworkopen.2025.19095. PMID 40627355